CLINICAL TRIAL: NCT05168163
Title: A Phase II Randomized Study of Atezolizumab Plus Multi-Kinase Inhibitor Versus Multi-Kinase Inhibitor Alone in Subjects With Unresectable, Advanced Hepatocellular Carcinoma Who Previously Received Atezolizumab Plus Bevacizumab
Brief Title: Atezolizumab in Combination With a Multi-Kinase Inhibitor for the Treatment of Unresectable, Locally Advanced, or Metastatic Liver Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-GI-2008; NCI-2021-12091 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-GI-2008 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2021-12-08; First posted 2021-12-23 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Hepatocellular Carcinoma; Metastatic Hepatocellular Carcinoma; Stage III Hepatocellular Carcinoma AJCC v8; Stage IIIA Hepatocellular Carcinoma AJCC v8; Stage IIIB Hepatocellular Carcinoma AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8; Stage IVA Hepatocellular Carcinoma AJCC v8; Stage IVB Hepatocellular Carcinoma AJCC v8; Unresectable Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; cabozantinib; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (atezolizumab, cabozantinib or lenvatinib) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on day 1 and cabozantinib PO QD or lenvatinib PO QD on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Atezolizumab; Drug: Cabozantinib; Drug: Lenvatinib
- Arm B (cabozantinib or lenvatinib) (Active Comparator): Patients receive cabozantinib PO QD or lenvatinib PO QD on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib; Drug: Lenvatinib

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
  Arms: Arm A (atezolizumab, cabozantinib or lenvatinib)
Drug: Cabozantinib — Given PO
Drug: Lenvatinib — Given PO
  Other Names: E7080; ER-203492-00; Multi-Kinase Inhibitor E7080

SUMMARY:
This phase II trial tests whether atezolizumab in combination with a multi-kinase inhibitor (cabozantinib or lenvatinib) compared to multi-kinase inhibitor alone in treating patients with liver cancer that cannot be removed by surgery (unresectable), has spread to has spread to nearby tissue or lymph nodes (locally advanced), or has spread to other places in the body (metastatic), for which the patient has received treatment in the past (previously treated). Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Cabozantinib and lenvatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving atezolizumab with cabozantinib or lenvatinib may kill more tumor cells in patients with liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the progression-free and overall survival in subjects with advanced hepatocellular carcinoma who previously progressed on atezolizumab/bevacizumab who are treated using atezolizumab plus a multi-kinase inhibitor compared to multi-kinase inhibitor alone.

SECONDARY OBJECTIVES:

I. To determine the overall response rate per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 response in subjects who are treated using atezolizumab plus a multi-kinase inhibitor compared to multi-kinase inhibitor alone.

II. To determine the duration of response in subjects who are treated using atezolizumab plus a multi-kinase inhibitor compared to multi-kinase inhibitor alone.

III. To determine the safety profile of adding atezolizumab to multi-kinase inhibitor in subjects who are treated using atezolizumab plus a multi-kinase inhibitor compared to multi-kinase inhibitor alone.

EXPLORATORY OBJECTIVE:

I. To explore for potential predictive biomarkers for response and resistance to anti-PD-L1 and/or multi-kinase inhibitor therapy in subject population.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive atezolizumab intravenously (IV) over 30-60 minutes on day 1 and cabozantinib orally (PO) once daily (QD) or lenvatinib PO QD on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive cabozantinib PO QD or lenvatinib PO QD on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed-up every 9 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent =< 28 days prior to randomization
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

  * NOTE: During the Active Monitoring Phase of a study (i.e., active treatment and clinical follow-up), participants must be willing to return to the consenting institution for follow-up
* Age >= 18 years
* Hepatocellular carcinoma (HCC) confirmed by histological/cytological diagnosis or clinically per the American Association for the Study of Liver Diseases (AASLD) or WASL 2018 criteria
* Locally advanced, metastatic and/or unresectable disease that is not amendable to curative treatment
* Previously progressed on atezolizumab in combination with bevacizumab as first line systemic therapy for advanced disease

  * NOTE: 2nd line patients only
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Child Pugh class A
* Documented virology status of hepatitis, as confirmed by screening hepatitis B virus (HBV) and hepatitis C virus (HCV) serology tests.

  * For subjects with active HBV, HBV deoxyribonucleic acid (DNA) < 500 IU/mL obtained ≤ =< 28 days prior to randomization, and anti-HBV treatment (per local standard of care; e.g., entecavir) for a minimum of 14 days prior to randomization and willingness to continue treatment for the length of the study
* At least one measurable untreated malignant lesion per RECIST v1.1. Subjects who previously received local therapy (e.g., ablation, percutaneous ethanol injection, trans-arterial embolization/chemo-embolization) are eligible provided the target lesion(s) have not been previously treated with local therapy or the target lesion(s) within the field of local therapy have subsequently progressed in accordance with RECIST v1.1
* Consent to using archival tumor tissues, if available

  * NOTE: Non-availability of tumor tissue does not exclude the subject.
* Willingness to provide mandatory blood specimens for correlative research
* Willingness to provide mandatory tissue specimens for correlative research for the first 10 patients per arm (Mayo Clinic Rochester and Mayo Clinic Arizona ONLY)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (1500/uL) without granulocyte colony-stimulating factor support (obtained =< 28 days prior to randomization)
* Lymphocyte count >= 0.5 x 10^9/L (500/uL) (obtained =< 28 days prior to randomization)
* Platelet count >= 75 x 10^9/L (75,000/uL) (obtained =< 28 days prior to randomization)
* Hemoglobin >= 90 g/L (9 g/dL) (obtained =< 28 days prior to randomization)

  * Subjects may be transfused to meet this criterion
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) =< 5 x upper limit of normal (ULN) (obtained =< 28 days prior to randomization)
* Total bilirubin =< 3 x ULN (obtained =< 28 days prior to randomization)
* Serum albumin >= 30 g/L (3.0 g/dL) (obtained =< 28 days prior to randomization)
* For subjects not receiving therapeutic anticoagulation: international normalized ratio (INR) or partial thromboplastin time (aPTT) =< 1.5 × ULN (obtained =< 28 days prior to randomization)
* Serum creatinine =< 2 x ULN or creatinine clearance >= 30 mL/min (calculated using the Cockcroft-Gault formula) (obtained =< 28 days prior to randomization)
* Negative pregnancy test done =< 14 days prior to randomization, for women of childbearing potential only

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Resolution of any acute, clinically significant treatment-related toxicity from prior therapy to grade =< 1 prior to randomization, with the exception of alopecia and peripheral sensory neuropathy.
* Subjects of childbearing potential agree to use two forms of medically approved contraception while taking the study drug and for at least 5 months after the last dose of atezolizumab or multi-kinase inhibitor. Subjects with partners of childbearing potential agree to use condoms, even after vasectomy, to avoid potential drug exposure to partner during study drug and for 5 months following the last dose of study drug
* Ability to take oral medications

Exclusion Criteria:

* Known diagnosis of fibrolamellar carcinoma, sarcomatoid carcinoma or mixed hepatocellular cholangiocarcinoma
* Prior multi-kinase inhibitor treatment for advanced disease (e.g., cabozantinib, lenvatinib, sorafenib, regorafenib)

  * NOTE: Use of multi-kinase inhibitor(s) for adjuvant or as part of loco-regional therapies is allowed as long as the therapy was completed >= 6 months prior to randomization
* Any of the following prior therapies:

  * Major surgery =< 4 weeks prior to randomization; Minor surgery =< 7 days prior to randomization (e.g., simple excision, tooth extraction, insertion of central lines/Mediport). Subjects with clinically relevant complications from prior surgery are not eligible
  * Any anti-cancer agent =< 2 weeks prior to randomization
  * Radiation therapy =< 4 weeks (1 week for palliative radiation for bone metastases and/or for pain control) or radionuclide treatment (e.g., I-131 or Y-90) =< 6 weeks prior to randomization
* Treatment with investigational therapy =< 28 days prior to randomization
* Known brain or leptomeningeal metastasis
* Known co-infection of HBV and HCV. Subjects with a history of HCV infection but who are negative for HCV ribonucleic acid (RNA) by polymerase chain reaction (PCR) will be considered non-infected with HCV
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis with the following exceptions:

  * Subjects with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study
  * Subjects with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
  * Subjects with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., subjects with psoriatic arthritis are excluded) are eligible for the study provided all of the following conditions are met:

    * Rash must cover < 10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan

  * NOTE: History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the subject at high risk from treatment complication
* Treatment with a live, attenuated vaccine =< 4 weeks prior to randomization, or anticipation of need for such a vaccine during atezolizumab treatment or =< 5 months after the last dose of atezolizumab
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Subjects with untreated or incompletely treated esophageal/gastric varices with bleeding or high risk for bleeding. Subjects treated with adequate endoscopic therapy (according to local institutional standards) without any episodes of recurrent gastrointestinal bleeding requiring transfusion or hospitalization for > 28 days prior to randomization are eligible
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) =< 4 weeks or 5 drug elimination half-lives (whichever is longer) prior to randomization
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies

  * Note: Prior treatment with atezolizumab is permitted
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF alpha agents) =< 2 weeks prior to randomization, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  * Subjects who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study
  * Subjects who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible
* For subjects who are to receive cabozantinib: Treatment with strong inducers and/or strong inhibitors of CYP3A4 =< 14 days prior to randomization, including rifampin (and its analogues) or St. John's wort. See https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers for lists of known strong inhibitors and strong inducers of CYP3A4
* Active tuberculosis
* Other uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders including:

    * Symptomatic congestive heart failure, unstable angina, or serious cardiac arrythmias
    * Uncontrolled hypertensions defined as sustained blood pressure (BP) > 150 mmHg systolic BP, or > 100 mmHg diastolic BP despite optimal antihypertensive treatment
    * Stroke (including transient ischemic attack), myocardial infarction, or other ischemic event =< 3 months prior to randomization.
    * Unstable arrythmia
    * Thromboembolic event =< 3 months prior to randomization. Subjects with thromboses of portal/hepatic vasculature attributed to underlying liver disease and/or liver tumor are eligible.
  * Active bacterial infection requiring systemic treatment. Subjects on prophylactic antibiotics are eligible.
  * Known human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS) related illness. Subjects with known HIV but without clinical evidence of an immunocompromised state and receiving anti-retroviral therapy are eligible
  * Prior allogenic stem cell or solid organ transplantation
  * Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)

    * Subjects with indwelling catheters (e.g., PleurX) are allowed.
  * Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
  * Uncontrolled tumor-related pain

    * Patients requiring pain medication must be on a stable regimen at the time of randomization
    * Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to randomization. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.
    * Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to randomization
* Other malignancy(ies) =< 5 years prior to randomization except adequately treated non-melanotic skin cancer, carcinoma-in-situ of the cervix, localized prostate cancer, ductal carcinoma in situ or stage I uterine cancer
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within at least 5 months after the last dose of study medication
* Uncontrolled hepatic encephalopathy occurring =< 6 weeks prior to randomization NOTE: Patients with =< grade 2 encephalopathy =< 6 weeks prior to randomization are eligible and supportive measures such as lactulose and antibiotics are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization to death from any cause, assessed up to 3 years
  The final analysis for OS will be conducted when 84 OS events are observed, approximately 36 months after first subject in and will be evaluated with a one-sided p-value from stratified log-rank test.
Progression-free survival (PFS) | From randomization to first documentation of disease progression (per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) or death, assessed up to 2 years
  PFS analysis will be conducted when 89 PFS events are observed. The one-sided p-value from stratified log-rank test will be used for decision making.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  Objective response is defined as either a complete response (CR) or partial response (PR) (as defined by the RECIST 1.1). ORR will be calculated by the number of subjects experience objective response divided by the number of evaluable subjects in each arm. Confidence intervals for the ORR will be calculated using a normal approximation and the corresponding 95% confidence interval will be reported.
Duration of response | Up to 2 years
  For subjects who experience a CR or PR, duration of response is defined as the time from the date of first response (CR or PR) to progression or death, whichever is earliest. Median duration for each arm and corresponding 95% confidence interval, calculated using Kaplan-Meier method and Brookmeyer-Crowley, will be reported.
Incidence of adverse events (AEs) | Up to 30 days after last dose
  Common Terminology Criteria for Adverse Events (CTCAE) AEs will be recorded for each subject. The overall adverse event rates for grade 3 or higher AEs will be reported by arm.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Wee Ma, Principal Investigator — Academic and Community Cancer Research United
Locations (16):
- United States (16):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Cleveland Clinic Weston Florida, Weston, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle Cancer Center NCI Community Oncology Research Program, Urbana, Illinois
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Froedtert and the Medical College of Wisconsin LAPS, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin